CLINICAL TRIAL: NCT00267098
Title: Biventricular Versus Right Ventricular Pacing in Heart Failure Patients With Atrioventricular Block (BLOCK HF)
Acronym: BLOCK HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Atrioventricular Block; Heart Diseases
Keywords: Atrioventricular block; Cardiac Resynchronization Therapy; Pacemaker; Defibrillator; NYHA Class I, II or III Heart failure
MeSH Terms: conditions — Atrioventricular Block; Heart Diseases | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biventricular pacing (Experimental)
  Interventions: Device: Cardiac Resynchronization Therapy (CRT)
- Right ventricular pacing (Active Comparator)
  Interventions: Device: Cardiac Resynchronization Therapy (CRT)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (CRT) — Biventricular pacing
  Other Names: Medtronic CRT-P; Medtronic CRT-D
  Arms: Biventricular pacing
Device: Cardiac Resynchronization Therapy (CRT) — Right ventricular pacing
  Other Names: Medtronic CRT-P; Medtronic CRT-D
  Arms: Right ventricular pacing

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heartbeat, sometimes a pacemaker is used to control the rate and rhythm of the heartbeat. In this trial, the researchers will test if pacing both the left and right lower half of the heart (ventricles) will:

* decrease the number of hospital and clinic visits due to heart failure symptoms
* extend life
* delay heart failure symptoms as compared to those who are paced in only one ventricle (the right ventricle)

ELIGIBILITY:
Inclusion Criteria:

* Subject has standard class I or class IIa indication for pacemaker implantation in accordance with ACC/AHA/HRS guidelines
* Subjects diagnosed with atrioventricular (AV) block. An AV block is a disturbance when the heart's natural pacemaker sends a message from the atrium (top part of heart) to the ventricle (bottom part of heart) and the message is partially or totally blocked
* Subject is receiving first time implant
* Subjects with heart failure but no symptoms of it (New York Heart Association [NYHA] Class I), or subjects with mild heart failure that only sometimes interferes with their daily activities (NYHA Class II), or subjects with heart failure that severely limits daily activities (NYHA Class III)
* Subjects with documented reduced heart pumping function (left ventricular ejection fraction ≤ 50%) within past 90 days
* Subject is at least 18 years old
* Subject or authorized legal guardian or representative has signed and dated the Informed Consent
* Subject is able to receive a pectoral implant
* Subject is expected to remain available for follow-up visits at the study center
* Subject is willing and able to comply with the protocol

Exclusion Criteria:

* Subject has ever had a previous or has an existing device implant
* Subjects with some forms of chest pain or myocardial infarction (heart attack) within the past 30 days
* Subjects with coronary bypass within the past 30 days
* Subjects with stent within the past 30 days
* Subjects with valve repair or replacement within the past 6 months or is indicated for repair or replacement
* Subjects with a mechanical right heart valve
* Subject is indicated for a biventricular pacing device (CRT-P or CRT-D devices)
* Subject is enrolled in a concurrent study which may confound the results of this study (co-enrollment in any concurrent clinical study requires approval of the study manager)
* Subject is pregnant, or of child bearing potential and not on a reliable form of birth control
* Subjects with a previous heart transplant
* Subjects has been classified as NHYA Functional Class IV within prior 90 days (subjects with severe heart failure and should always be resting)
* Subject, legal guardian or authorized representative is unable or unwilling to cooperate or give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Actual)
Dates: Start 2003-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne B. Curtis, MD, FHRS, FACC, Principal Investigator — University at Buffalo, NY
Locations (54):
- United States (51):
  - Anchorage, Alaska
  - Peoria, Arizona
  - Little Rock, Arkansas
  - Glendale, California
  - Long Beach, California
  - Colorado Springs, Colorado
  - Hollywood, Florida
  - Jacksonville, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Park Ridge, Illinois
  - Rockford, Illinois
  - Davenport, Iowa
  - Lexington, Kentucky
  - Lacombe, Louisiana
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Petoskey, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Saint Louis Park, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Camden, New Jersey
  - Hackensack, New Jersey
  - Ridgewood, New Jersey
  - Bay Shore, New York
  - Rochester, New York
  - Syracuse, New York
  - West Islip, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Danville, Pennsylvania
  - Doylestown, Pennsylvania
  - Ephrata, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wynnewood, Pennsylvania
  - Wyomissing, Pennsylvania
  - Providence, Rhode Island
  - Kingsport, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Spokane, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Canada (3):
  - Kitchener, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Fudim M, Dalgaard F, Friedman DJ, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Ali-Ahmed F, Tang A, Olivas-Martinez A, Inoue LYT, Al-Khatib SM, Sanders GD. Comorbidities and clinical response to cardiac resynchronization therapy: Patient-level meta-analysis from eight clinical trials. Eur J Heart Fail. 2024 Apr;26(4):1039-1046. doi: 10.1002/ejhf.3029. Epub 2023 Sep 15. PMID 37671601
- [Derived] Friedman DJ, Al-Khatib SM, Dalgaard F, Fudim M, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Tang AS, Ali-Ahmed F, Olivas-Martinez A, Inoue LYT, Sanders GD. Cardiac Resynchronization Therapy Improves Outcomes in Patients With Intraventricular Conduction Delay But Not Right Bundle Branch Block: A Patient-Level Meta-Analysis of Randomized Controlled Trials. Circulation. 2023 Mar 7;147(10):812-823. doi: 10.1161/CIRCULATIONAHA.122.062124. Epub 2023 Jan 26. PMID 36700426
- [Derived] Curtis AB, Worley SJ, Chung ES, Li P, Christman SA, St John Sutton M. Improvement in Clinical Outcomes With Biventricular Versus Right Ventricular Pacing: The BLOCK HF Study. J Am Coll Cardiol. 2016 May 10;67(18):2148-2157. doi: 10.1016/j.jacc.2016.02.051. PMID 27151347
- [Derived] St John Sutton M, Plappert T, Adamson PB, Li P, Christman SA, Chung ES, Curtis AB. Left Ventricular Reverse Remodeling With Biventricular Versus Right Ventricular Pacing in Patients With Atrioventricular Block and Heart Failure in the BLOCK HF Trial. Circ Heart Fail. 2015 May;8(3):510-8. doi: 10.1161/CIRCHEARTFAILURE.114.001626. Epub 2015 Feb 19. PMID 25697851
- [Derived] Curtis AB, Worley SJ, Adamson PB, Chung ES, Niazi I, Sherfesee L, Shinn T, Sutton MS; Biventricular versus Right Ventricular Pacing in Heart Failure Patients with Atrioventricular Block (BLOCK HF) Trial Investigators. Biventricular pacing for atrioventricular block and systolic dysfunction. N Engl J Med. 2013 Apr 25;368(17):1585-93. doi: 10.1056/NEJMoa1210356. PMID 23614585

RESULTS

PARTICIPANT FLOW:
Groups:
- No Implant Attempt: Subjects who did not undergo an implant attempt of a CRT-P or CRT-D device and were not randomized
- Unsuccessful Implants: Subjects who underwent an implant attempt of a CRT-P or CRT-D device but were not successfully implanted
- CRT-P: Biventricular Pacing Arm: Subjects who were implanted with a CRT-P device and randomized to receive biventricular pacing
- CRT-P: Right Ventricular Pacing Arm: Subjects who were implanted with a CRT-P device and randomized to receive right ventricular pacing
- CRT-P: Not Randomized: Subjects successfully implanted with a CRT-P device who were not randomized
- CRT-D: Biventricular Pacing Arm: Subjects implanted with a CRT-D device and randomized to receive biventricular pacing
- CRT-D: Right Ventricular Pacing Arm: Subjects implanted with a CRT-D device and randomized to receive right ventricular pacing.
- CRT-D: Not Randomized: Subjects successfully implanted with a CRT-D device who were not randomized
Period: Overall Study
Arm/Group | No Implant Attempt | Unsuccessful Implants | CRT-P: Biventricular Pacing Arm | CRT-P: Right Ventricular Pacing Arm | CRT-P: Not Randomized | CRT-D: Biventricular Pacing Arm | CRT-D: Right Ventricular Pacing Arm | CRT-D: Not Randomized
Started | 109 | 51 | 243 | 241 | 47 | 106 | 101 | 20
Completed | 0 | 0 | 149 | 135 | 10 | 66 | 55 | 5
Not Completed | 109 | 51 | 94 | 106 | 37 | 40 | 46 | 15
Not completed — Death | 0 | 0 | 57 | 66 | 14 | 23 | 28 | 9
Not completed — Lost to Follow-up | 0 | 0 | 6 | 5 | 2 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 0 | 24 | 21 | 12 | 9 | 12 | 5
Not completed — Physician Decision | 5 | 0 | 7 | 11 | 5 | 4 | 3 | 0
Not completed — Inclusion/Exclusion Criteria Not Met | 96 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Unsuccessful Implant Exit Per Protocol | 0 | 51 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site closure | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Explanted Medtronic device | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non-Medtronic LV Lead Implanted | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Subject listed for heart transplant | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor withdrew subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Implant Attempt | Unsuccessful Implants | CRT-P: Biventricular Pacing Arm | CRT-P: Right Ventricular Pacing Arm | CRT-P: Not Randomized | CRT-D: Biventricular Pacing Arm | CRT-D: Right Ventricular Pacing Arm | CRT-D: Not Randomized | Total
Number analyzed (Participants) | 109 | 51 | 243 | 241 | 47 | 106 | 101 | 20 | 918
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (12.6) | 71.1 (11.2) | 74.4 (10.2) | 73.8 (10.8) | 79.3 (7.6) | 72.0 (9.3) | 71.0 (10.0) | 74.0 (9.1) | 73.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 14 | 62 | 73 | 18 | 19 | 20 | 4 | 239
  Male | 80 | 37 | 181 | 168 | 29 | 87 | 81 | 16 | 679
Race/Ethnicity, Customized [Number; unit: participants]
  Subject did not offer ethnicity | 6 | 2 | 6 | 5 | 1 | 4 | 3 | 0 | 27
  African American | 10 | 3 | 8 | 10 | 0 | 4 | 4 | 1 | 40
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Caucasian | 91 | 45 | 225 | 224 | 43 | 96 | 90 | 18 | 832
  Hispanic | 1 | 0 | 3 | 1 | 2 | 2 | 2 | 1 | 12
  Native American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 109 | 46 | 232 | 231 | 47 | 104 | 98 | 19 | 886
  Canada | 0 | 5 | 11 | 10 | 0 | 2 | 3 | 1 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mortality, Heart Failure-related Urgent Care Visits, or Significant Increase in Left Ventricular End Systolic Volume Index (LVESVI)
Description: Events include all-cause mortality, heart failure(HF)-related urgent care (a healthcare utilization visit involving intravenous(IV) therapy for heart failure) or significant increase(at least 15%) in LVESVI (a measure of the volume of a patient's left ventricle) from randomization to a later time point. Time from randomization until the subject experienced one of these events served as the outcome measure. LVESVI endpoints occurred primarily at those visits in which LVESVI measurements were required (6, 12, 18, 24 months). Because endpoints such as death or HF urgent care could occur at any time during follow-up, the subject's outcome measure could range from less than 1 month to 105 months (maximum follow-up duration). Primary endpoints and follow-up data occurring after a subject missed a required LVESVI measurement were excluded from the analysis and the table below. The counts reflect the number of subjects meeting each endpoint, and are not necessarily mutually exclusive.
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: Only randomized subjects in both device groups were included in the analysis of this endpoint, as the analysis was restricted to post-randomization data. Subjects in the "No Implant Attempt", "Unsuccessful Implants", "CRT-P: Not Randomized", and "CRT-D: Not Randomized" subgroups were excluded.
Measure: Number; unit: participants
Groups:
- Biventricular Pacing Arm: Subjects randomized to receive biventricular pacing
- Right Ventricular Pacing Arm: Subjects randomized to receive right ventricular pacing.
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Subjects Experiencing a Primary Endpoint | 160 | 191
  Subjects with an LVESVI Primary Endpoint | 93 | 136
  Subjects with an HF Urgent Care Primary Endpoint | 70 | 94
  Subjects who died | 55 | 66
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same rate of mortality, a heart failure urgent care visit, or significant increase in LVESVI as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a lower rate of this composite endpoint than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.9990, Posterior Distribution for HR — BLOCK HF is a Bayesian study;a p-value was not used. Instead, a posterior probability,representing the probability that patients with BiV pacing have lower risk of events than those with RV pacing, was calculated. A probability ≥0.95 was significant; The posterior distribution is the set of values the BiV to RV hazard ratio can take, and its likelihood of taking such values; Hazard Ratio (HR) = 0.729, 95% CI 2-sided [0.592 to 0.889] — The hazard ratio corresponds to the time until death, a HF urgent care event or visit in which the LVESVI endpoint was met. Data beyond missed LVESVI measurements were excluded. A 95% credible interval was used instead of a 95% confidence interval

2. Secondary Outcome: All-Cause Mortality
Description: The endpoint is the time to death from any cause. The rate of mortality, as measure by the hazard rate, in each randomization arm will be compared.
  This outcome includes all post-randomization deaths, whereas the reporting of the primary outcome excluded primary endpoints (including deaths) that occurred after the subject had missed a study-required echocardiogram (used to determine if the LVESVI primary endpoint was met).
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Subjects who died | 80 | 94
  Subjects who did not die | 269 | 248
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same rate of mortality as corresponding patients who receive right ventricular pacing; Test type: Superiority or Other; p = 0.865, Posterior Distribution for HR — BLOCK HF is a Bayesian study; thus p-values were not used. Instead, posterior probabilities, representing the probability that subjects with biventricular pacing have better outcomes, were calculated. A probability ≥ 0.95 was significant; The posterior distribution is the set of values the BiV to RV hazard ratio for death can take, and its likelihood of taking such values; Hazard Ratio (HR) = 0.843, 95% CI 2-sided [0.632 to 1.142] — Because BLOCK HF was a Bayesian study, a 95% credible interval was used in lieu of a 95% confidence interval. This interval reflects the set of values the Hazard Ratio can take with 95% posterior probability

3. Secondary Outcome: All-Cause Mortality or Heart Failure-related Hospitalization
Description: The endpoint will be a subject's time from randomization to either their first heart failure-related hospitalization, or death.
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Subjects who died or underwent HF hospitalization | 121 | 135
  Subjects who died | 80 | 94
  Subjects who underwent HF hospitalization | 79 | 92
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same rate of mortality or heart failure(HF)-related hospitalization as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a lower rate of death or first HF hospitalization than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.9785, Posterior Distribution for HR — BLOCK HF is a Bayesian study; a p-value was not used. Instead, a posterior probability, representing the probability that patients with BiV pacing have better outcomes than those with RV pacing, was calculated. A probability ≥0.95 was significant; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.781, 95% CI 2-sided [0.615 to 0.991] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: All-Cause Mortality or Significant Increase in Left Ventricular End Systolic Volume Index
Description: The endpoint will be the time from randomization to either death or a visit (6, 12, 18, 24 month or interim visit) in which the subject undergoes an echocardiogram and the measured left ventricular end systolic volume index (a measure of the size of the subject's left ventricle normalized over their body surface area) is at least 15% greater than the corresponding measured value at randomization.
  Only LVESVI endpoints/deaths and follow-up data occurring before a subject missed an LVESVI measurement (due to missed visit, echo not performed, etc.) were used in the analysis and included in the table below. The counts reflect the number of subjects meeting each endpoint, and are not mutually exclusive.
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Subjects who died or experienced LVESVI event | 131 | 171
  Subjects who died | 55 | 66
  Subjects who experienced LVESVI event | 93 | 136
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or II who receive biventricular pacing have the same rate of mortality or significant increase in LVESVI as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a lower rate of death or significant increase in LVESVI than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.9886, Posterior Distribution for HR — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.695, 95% CI 2-sided [0.558 to 0.866] — The hazard ratio corresponds to the time from randomization to death or a visit in which LVESVI endpoint was met. Data beyond missed LVESVI measurements were excluded. A 95% credible interval was used instead of a 95% confidence interval

5. Secondary Outcome: First Heart Failure Hospitalization
Description: The endpoint is the time from randomization to a subject's first heart failure (HF)-related hospitalization. For each randomization arm, the number of subjects who met the endpoint, experiencing at least one heart failure-related hospitalization post-randomization, are reported, as well as the number of randomized subjects who did not experience any HF hospitalizations post-randomization.
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Subjects experiencing a HF hospitalization | 79 | 92
  Subjects not experiencing a HF hospitalization | 270 | 250
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same rate of first heart failure(HF)-related hospitalization as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a lower rate of first HF hospitalization than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.9904, Posterior Distribution for HR — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.704, 95% CI 2-sided [0.522 to 0.947] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Days Hospitalized for Heart Failure
Description: For each subject the endpoint was the days hospitalized for heart failure per patient year, calculated as the total number of days the subject was hospitalized for heart failure divided by the subject's total follow-up time. Only post-randomization data were used.
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days hospitalized per patient year
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
Days hospitalized per patient year | 1.89 (9.52) | 2.63 (16.08)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same rate of days hospitalized for heart failure per year as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a lower rate of days hospitalized for HF than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.637, Difference in Average Ranks — [p-value comment as in outcome 3, analysis 1]; The subjects' individual rates of days hospitalized for HF were ranked, with lower ranks corresponding to fewer days hospitalized for HF; BiV - RV Difference in Average Rank = -1.8 — The posterior probability that the BiV - RV difference in average ranks was below 0 (denoting that the BiV arm had lower ranks than the RV arm, on average) was calculated

7. Secondary Outcome: Change in New York Heart Association Classification
Description: The endpoint is a subject's change in New York Heart Association Classification (a measure of the degree of heart failure a subject has on a 4 class scale, with NYHA I being the healthiest score and NYHA IV being the sickest score) from randomization to each of four time points: 6 months, 12 months, 18 months, and 24 months post-randomization. The change categories listed will be relative to randomization.
Time Frame: Randomization to 24 Months
Population: For each time point(e.g. 6 months), only subjects with NYHA assessed at both randomization and that time point were included in the analysis. Those who could not be analyzed at a time point(for reasons such as death, exit,missed visit,or NYHA not assessed at visit) are listed under the "Comparative data not available" category for that time point.
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  6 Months: Improved by 2 classes from randomization | 5 | 3
  6 Months: Improved by 1 class from randomization | 54 | 43
  6 Months: No change from randomization | 200 | 205
  6 Months: Worsened by 1 class from randomization | 52 | 41
  6 Months: Worsened by 2 classes from randomization | 1 | 1
  6 Months: Comparative data not available | 37 | 49
  12 Months:Improved by 2 classes from randomization | 4 | 5
  12 Months:Improved by 1 class from randomization | 54 | 34
  12 Months: No change from randomization | 172 | 172
  12 Months: Worsened by 1 class from randomization | 49 | 64
  12 Months:Worsened by 2 classes from randomization | 2 | 3
  12 Months: Comparative data not available | 68 | 64
  18 Months:Improved by 2 classes from randomization | 3 | 2
  18 Months: Improved by 1 class from randomization | 43 | 45
  18 Months: No change from randomization | 142 | 141
  18 Months: Worsened by 1 class from randomization | 50 | 56
  18 Months:Worsened by 2 classes from randomization | 4 | 6
  18 Months: Comparative data not available | 107 | 92
  24 Months:Improved by 2 classes from randomization | 2 | 3
  24 Months: Improved by 1 class from randomization | 35 | 36
  24 Months: No change from randomization | 135 | 126
  24 Months:Worsened by 1 class from randomization | 41 | 54
  24 Months:Worsened by 2 classes from randomization | 4 | 3
  24 Months: Comparative data not available | 132 | 120
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in NYHA classification from randomization to 6 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.591, Posterior Distribution for Average Rank — BLOCK HF is a Bayesian study; thus p-values were not used. Instead, a posterior probability, representing the probability that subjects with biventricular pacing have better outcomes at 6 months, was calculated. A probability ≥0.95 was significant; Subjects' Randomization - 6 month changes in NYHA classification were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.012 — Positive values reflect better outcomes over time in the BiV arm than the RV arm
Statistical Analysis 2: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in NYHA classification from randomization to 12 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.986, Posterior Distribution for Average Rank — BLOCK HF is a Bayesian study; thus p-values were not used. Instead, a posterior probability,representing the probability that subjects with biventricular pacing have better outcomes at 12 months, was calculated. A probability ≥0.95 was significant; Subjects' Randomization - 12 month changes in NYHA classification were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.126 — Positive values reflect better outcomes over time in the BiV arm than the RV arm
Statistical Analysis 3: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in NYHA classification from randomization to 18 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.726, Posterior Distribution for Average Rank — [p-value comment as in outcome 7, analysis 2]; Subjects' Randomization - 18 month changes in NYHA classification were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.039 — Positive values reflect better outcomes over time in the BiV arm than the RV arm
Statistical Analysis 4: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in NYHA classification from randomization to 24 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.701, Posterior Distribution for Average Rank — BLOCK HF is a Bayesian study; thus p-values were not used. Instead, a posterior probability,representing the probability that subjects with biventricular pacing have better outcomes at 24 months, was calculated. A probability ≥0.95 was significant; Subjects' Randomization - 24 month changes in NYHA classification were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.035 — Positive values reflect better outcomes over time in the BiV arm than the RV arm

8. Secondary Outcome: Change in Heart Failure Stage
Description: The endpoint is a subject's change in Heart Failure Stage (a measure of the degree of heart failure a subject has on a 4 stage scale (A, B, C, D), with Class A being the healthiest score and Class D being the sickest score) from randomization to each of four time points: 6 months, 12 months, 18 months, and 24 months.
Time Frame: Randomization to 24 Months
Population: For each time point(e.g. 6 months), only subjects with HF Stage assessed at randomization and that time point were included in the analysis. Those who could not be analyzed at a time point(for reasons such as death, exit,missed visit,or HF Stage not assessed) are listed under the "Comparative data not available" category for that time point.
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  6 Months: Improved by 2 stages since randomization | 1 | 0
  6 Months: Improved by 1 stage since randomization | 11 | 5
  6 Months: No change from randomization | 296 | 274
  6 Months: Worsened by 1 stage since randomization | 2 | 14
  6 Months: Worsened by 2 stages since randomization | 1 | 0
  6 Months: Comparative data not available | 38 | 49
  12 Months:Improved by 2 stages since randomization | 0 | 0
  12 Months:Improved by 1 stage since randomization | 7 | 8
  12 Months: No change since randomization | 258 | 244
  12 Months: Worsened by 1 stage since randomization | 15 | 23
  12 Months:Worsened by 2 stages since randomization | 1 | 1
  12 Months: Comparative data not available | 68 | 66
  18 Months:Improved by 2 stages since randomization | 0 | 0
  18 Months:Improved by 1 stage since randomization | 4 | 5
  18 Months: No change since randomization | 222 | 225
  18 Months:Worsened by 1 stage since randomization | 16 | 18
  18 Months:Worsened by 2 stages since randomization | 0 | 1
  18 Months: Comparative data not available | 107 | 93
  24 Months:Improved by 2 stages since randomization | 0 | 0
  24 Months: Improved by 1 stage since randomization | 4 | 6
  24 Months: No change since randomization | 196 | 197
  24 Months:Worsened by 1 stage since randomization | 16 | 19
  24 Months:Worsened by 2 stages since randomization | 1 | 0
  24 Months: Comparative data not available | 132 | 120
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in HF stage from randomization to 6 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.534, Posterior Distribution for Average Rank — [p-value comment as in outcome 7, analysis 1]; Subjects' Randomization - 6 month change in HF Stage were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.002 — Positive values reflect better outcomes over time in the BiV arm than the RV arm
Statistical Analysis 2: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' change in HF stage from randomization to 12 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.825, Posterior Distribution for Average Rank — [p-value comment as in outcome 7, analysis 2]; Subjects' Randomization - 12 month changes in HF Stage were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.026 — Positive values reflect better outcomes over time in the BiV arm than the RV arm
Statistical Analysis 3: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in HF stage from randomization to 18 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.651, Posterior Distribution for Average Rank — BLOCK HF is a Bayesian study; thus p-values were not used. Instead, a posterior probability,representing the probability that subjects with biventricular pacing have better outcomes at 18 months, was calculated. A probability ≥0.95 was significant; Subjects' Randomization - 18 month changes in HF Stage were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = 0.010 — Positive values denote that the BiV arm had better outcomes over time than the RV arm
Statistical Analysis 4: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; Subjects' changes in HF stage from randomization to 24 months were determined. The null hypothesis was that the average change among patients with biventricular pacing is equal to that of patients with right ventricular pacing; Test type: Superiority or Other; p = 0.425, Posterior Distribution for Average Rank — [p-value comment as in outcome 7, analysis 4]; Subjects' Randomization - 24 month changes in HF Stage were ranked. The BiV - RV difference in average rank was analyzed; BiV - RV Difference in Average Rank = -0.006 — Positive values denote better outcomes over time in the BiV arm than the RV arm

9. Secondary Outcome: Change in Cardiovascular Medications
Description: The endpoints are what classes of drugs (e.g. Beta blockers, Diuretics, Nitrates, etc.) each subject was on at the time of scheduled visits (e.g Randomization, 6 months, 12 months, etc.)
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Population: Because indications for defibrillation devices like CRT-Ds are defined by characteristics that relate to medication guidelines, medication results are presented separately for each device group. Medications were assessed only for subjects who completed visits (denoted as "Subjects with Medications Assessed").
Measure: Number; unit: participants
Groups:
- CRT-P: Biventricular Pacing Arm: Subjects implanted with a CRT-P device and randomized to receive biventricular pacing
- CRT-P: Right Ventricular Pacing Arm; CRT-D: Right Ventricular Pacing Arm: Subjects implanted with a CRT-D device and randomized to receive right ventricular pacing.
Arm/Group | CRT-P: Biventricular Pacing Arm | CRT-P: Right Ventricular Pacing Arm | CRT-D: Biventricular Pacing Arm | CRT-D: Right Ventricular Pacing Arm
Number analyzed (Participants) | 243 | 241 | 106 | 101
participants
  Randomization: Subjects on ACE-Inhibitors/ARBs | 173 | 179 | 93 | 84
  Randomization: Subjects on Beta Blockers | 186 | 191 | 98 | 93
  Randomization: Subjects on Vasodilators/Nitrates | 53 | 44 | 31 | 20
  Randomization: Subjects on Aldosterone Antagonists | 33 | 25 | 19 | 25
  Randomization: Subjects on Diuretics | 156 | 158 | 74 | 74
  6 Months: Subjects with Medications Assessed | 226 | 207 | 94 | 89
  6 Months: Subjects on ACE-Inhibitors/ARBs | 162 | 152 | 77 | 73
  6 Months: Subjects on Beta Blockers | 175 | 171 | 87 | 79
  6 Months: Subjects on Vasodilators/Nitrates | 46 | 42 | 24 | 12
  6 Months: Subjects on Aldosterone Antagonists | 31 | 21 | 20 | 25
  6 Months: Subjects on Diuretics | 148 | 137 | 66 | 70
  12 Months: Subjects with Medications Assessed | 205 | 200 | 83 | 81
  12 Months: Subjects on ACE-Inhibitors/ARBs | 147 | 151 | 72 | 70
  12 Months: Subjects on Beta Blockers | 158 | 170 | 79 | 75
  12 Months: Subjects on Vasodilators/Nitrates | 45 | 43 | 22 | 13
  12 Months: Subjects on Aldosterone Antagonists | 23 | 20 | 13 | 21
  12 Months: Subjects on Diuretics | 133 | 131 | 57 | 60
  18 Months: Subjects with Medications Assessed | 169 | 181 | 78 | 72
  18 Months: Subjects on ACE-Inhibitors/ARBs | 121 | 137 | 62 | 58
  18 Months: Subjects on Beta Blockers | 134 | 152 | 75 | 63
  18 Months: Subjects on Vasodilators/Nitrates | 36 | 44 | 22 | 11
  18 Months: Subjects on Aldosterone Antagonists | 16 | 21 | 9 | 20
  18 Months: Subjects on Diuretics | 111 | 125 | 51 | 59
  24 Months: Subjects with Medications Assessed | 152 | 157 | 69 | 67
  24 Months: Subjects on ACE-Inhibitors/ARBs | 114 | 119 | 58 | 56
  24 Months: Subjects on Beta Blockers | 118 | 133 | 65 | 63
  24 Months: Subjects on Vasodilators/Nitrates | 28 | 37 | 23 | 10
  24 Months: Subjects on Aldosterone Antagonists | 18 | 15 | 13 | 18
  24 Months: Subjects on Diuretics | 97 | 104 | 47 | 56
  30 Months: Subjects with Medications Assessed | 130 | 131 | 53 | 57
  30 Months: Subjects on ACE-Inhibitors/ARBs | 92 | 102 | 42 | 47
  30 Months: Subjects on Beta Blockers | 104 | 114 | 51 | 56
  30 Months: Subjects on Vasodilators/Nitrates | 23 | 28 | 16 | 11
  30 Months: Subjects on Aldosterone Antagonists | 14 | 14 | 10 | 15
  30 Months: Subjects on Diuretics | 82 | 90 | 36 | 50
  36 Months: Subjects with Medications Assessed | 109 | 112 | 42 | 44
  36 Months: Subjects on ACE-Inhibitors/ARBs | 76 | 85 | 30 | 37
  36 Months: Subjects on Beta Blockers | 86 | 97 | 41 | 44
  36 Months: Subjects on Vasodilators/Nitrates | 21 | 24 | 14 | 9
  36 Months: Subjects on Aldosterone Antagonists | 10 | 19 | 8 | 10
  36 Months: Subjects on Diuretics | 69 | 79 | 34 | 37
  42 Months: Subjects with Medications Assessed | 94 | 99 | 38 | 42
  42 Months: Subjects on ACE-Inhibitors/ARBs | 69 | 73 | 27 | 35
  42 Months: Subjects on Beta Blockers | 75 | 86 | 35 | 42
  42 Months: Subjects on Vasodilators/Nitrates | 15 | 22 | 12 | 10
  42 Months: Subjects on Aldosterone Antagonists | 8 | 13 | 9 | 12
  42 Months: Subjects on Diuretics | 57 | 71 | 31 | 39

10. Secondary Outcome: Frequency of Adverse Events Post-randomization
Description: Adverse events that subjects experienced after they were randomized were compared between arms with regard to several categories such as heart failure (HF)-relatedness, relatedness to the implant procedure, and relatedness to the implanted system, including individual components such as the left ventricular (LV) lead and the CRT-P or CRT-D generator.
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Measure: Number; unit: participants
Arm/Group | CRT-P: Biventricular Pacing Arm | CRT-P: Right Ventricular Pacing Arm | CRT-D: Biventricular Pacing Arm | CRT-D: Right Ventricular Pacing Arm
Number analyzed (Participants) | 243 | 241 | 106 | 101
participants
  Subjects with procedure-related AE(s) | 37 | 7 | 7 | 2
  Subjects with system-related AE(s) | 56 | 31 | 47 | 24
  Subjects with LV lead-related AE(s) | 40 | 12 | 14 | 4
  Subjects with CRT-P/CRT-D related AE(s) | 12 | 17 | 36 | 18
  Subjects with HF-related AE(s) | 73 | 106 | 45 | 47

11. Secondary Outcome: Cardiovascular-related Healthcare Utilizations
Description: Cardiovascular-related healthcare utilizations (HCUs), such as hospitalizations, Emergency Department visits, urgent care visits, and clinic visits that subjects experienced after being randomized were summarized for each randomization arm
Time Frame: Participants were followed for the duration of the study, an average of 39.8 months post-randomization.
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Subjects with a post-randomization CV HCU | 264 | 263
  Subjects with post-randomization hospitalization | 164 | 162
  Subjects with post-randomization ED visit | 118 | 128
  Subjects with post-randomization urgent care visit | 12 | 12
  Subjects with post-randomization clinic visit | 214 | 220

12. Secondary Outcome: Change in Quality of Life at 6 Months
Description: The endpoint will be a subject's change in Quality of Life score from randomization to 6 months. The Quality of Life score at a time point is calculated using the Minnesota Living with Heart Failure Questionnaire, which consists of 21 questions each on a 6 point scale from 0 to 5. The 21 scores are added up and the final score, ranging from 0 (best) to 105 (worst) is the subject's quality of life score. For each subject the measure will be the randomization visit - 6 month difference in QOL score, with positive values denoting a reduction in score and improvement in Quality of Life.
  Subjects with missing QOL scores at one or both time points were excluded from analysis, and so the number of subjects analyzed for this outcome was a subset of the number of randomized subjects.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 304 | 289
units on a scale | 5 (20.3) | 0.3 (19.4)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in QOL score from randomization to 6 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a greater reduction (and thus improvement) in QOL score at 6 months than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.9976, Posterior Probability of Mean QOL Change — [p-value comment as in outcome 3, analysis 1]; The posterior distribution for the BiV - RV difference in mean QOL score improvement from randomization to 6 months was determined; Mean Difference (Final Values) = 4.7

13. Secondary Outcome: Change in Quality of Life at 12 Months
Description: The endpoint will be a subject's change in Quality of Life score from randomization to 12 months. The Quality of Life score at a time point is calculated using the Minnesota Living with Heart Failure Questionnaire, which consists of 21 questions each on a 6 point scale from 0 to 5. The 21 scores are added up and the final score, ranging from 0 (best) to 105 (worst) is the subject's quality of life score. For each subject the measure will be the randomization visit - 12 month difference in QOL score, with positive values denoting a reduction in score and improvement in Quality of Life.
  Subjects with missing QOL scores at one or both time points were excluded from analysis, and so the number of subjects analyzed for this outcome was a subset of the number of randomized subjects.
Time Frame: Randomization to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 274 | 273
units on a scale | 3.9 (20.1) | 0.9 (18.9)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in QOL score from randomization to 12 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a greater reduction (and thus improvement) in QOL score at 12 months than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.9641, Posterior Probability of Mean QOL Change — [p-value comment as in outcome 3, analysis 1]; The posterior distribution for the BiV - RV difference in mean QOL score improvement from randomization to 12 months was determined; Mean Difference (Final Values) = 3.0

14. Secondary Outcome: Change in Quality of Life at 18 Months
Description: The endpoint will be a subject's change in Quality of Life score from randomization to 18 months. The Quality of Life score at a time point is calculated using the Minnesota Living with Heart Failure Questionnaire, which consists of 21 questions each on a 6 point scale from 0 to 5. The 21 scores are added up and the final score, ranging from 0 (best) to 105 (worst) is the subject's quality of life score. For each subject the measure will be the randomization visit - 18 month difference in QOL score, with positive values denoting a reduction in score and improvement in Quality of Life.
  Subjects with missing QOL scores at one or both time points were excluded from analysis, and so the number of subjects analyzed for this outcome was a subset of the number of randomized subjects.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 237 | 244
units on a scale | 2.3 (20.5) | 0.5 (18.1)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in QOL score from randomization to 18 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a greater reduction (and thus improvement) in QOL score at 18 months than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.8416, Posterior Probability of Mean QOL Change — [p-value comment as in outcome 3, analysis 1]; The parameter of interest was the BiV - RV difference in mean QOL change from randomization to 18 months; Mean Difference (Final Values) = 1.8

15. Secondary Outcome: Change in Quality of Life at 24 Months
Description: The endpoint will be a subject's change in Quality of Life score from randomization to 24 months. The Quality of Life score at a time point is calculated using the Minnesota Living with Heart Failure Questionnaire, which consists of 21 questions each on a 6 point scale from 0 to 5. The 21 scores are added up and the final score, ranging from 0 (best) to 105 (worst) is the subject's quality of life score. For each subject the measure will be the randomization visit - 24 month difference in QOL score, with positive values denoting a reduction in score and improvement in Quality of Life.
  Subjects with missing QOL scores at one or both time points were excluded from analysis, and so the number of subjects analyzed for this outcome was a subset of the number of randomized subjects.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 214 | 218
units on a scale | 2.6 (20.5) | 1.5 (18.8)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in QOL score from randomization to 24 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a greater reduction (and thus improvement) in QOL score at 24 months than patients with right ventricular pacing; Test type: Superiority or Other; p = 0.7270, Posterior Probability of Mean QOL Change — [p-value comment as in outcome 3, analysis 1]; The posterior distribution for the BiV - RV difference in mean QOL score improvement from randomization to 24 months was determined; Mean Difference (Final Values) = 1.1

16. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Randomization to 6 Months
Description: The endpoint will be a subject's change in LV Ejection Fraction (a measure of the percentage of blood ejected from the left ventricle of the heart with each contraction). A normal range is 55% to 70%. For each subject the measure will be the 6 month - randomization visit difference in LVEF value.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 282 | 273
percentage | 3.0 (8.4) | -0.3 (8.9)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEF from randomization to 6 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEF from randomization to 6 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead, a posterior distribution representing the set of possible values for the BiV - RV difference in improvement in LVEF through 6 months was used; Posterior BiV - RV Mean Difference = 3.334, 95% CI 2-sided [1.886 to 4.815] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEF change through 6 months

17. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Randomization to 12 Months
Description: The endpoint will be a subject's change in LV Ejection Fraction (a measure of the percentage of blood ejected from the left ventricle of the heart with each contraction). A normal range is 55% to 70%. For each subject the measure will be the 12 month - randomization visit difference in LVEF value.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 263 | 260
percentage | 2.7 (9.3) | -0.5 (9.4)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEF from randomization to 12 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEF from randomization to 12 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead, a posterior distribution representing the set of possible values for the BiV - RV difference in improvement in LVEF through 12 months was used; Posterior BiV - RV Mean Difference = 3.232, 95% CI 2-sided [1.618 to 4.839] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEF change through 12 months

18. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Randomization to 18 Months
Description: The endpoint will be a subject's change in LV Ejection Fraction (a measure of the percentage of blood ejected from the left ventricle of the heart with each contraction). A normal range is 55% to 70%. For each subject the measure will be the 18 month - randomization visit difference in LVEF value.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 223 | 226
percentage | 2.7 (9.5) | 0.4 (10.1)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEF from randomization to 18 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEF from randomization to 18 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead, a posterior distribution representing the set of possible values for the BiV - RV difference in improvement in LVEF at 18 months was used; Posterior BiV - RV Mean Difference = 2.240, 95% CI 2-sided [0.419 to 4.066] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEF change through 18 months

19. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Randomization to 24 Months
Description: The endpoint will be a subject's change in LV Ejection Fraction (a measure of the percentage of blood ejected from the left ventricle of the heart with each contraction). A normal range is 55% to 70%. For each subject the measure will be the 24 month - randomization visit difference in LVEF value.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 192 | 205
percentage | 2.0 (9.6) | -1.6 (10.5)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEF from randomization to 24 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEF from randomization to 24 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead, a posterior distribution representing the set of possible values for the BiV - RV difference in improvement in LVEF through 24 months was used; Posterior BiV - RV Mean Difference = 3.623, 95% CI 2-sided [1.623 to 5.604] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEF change through 24 months

20. Secondary Outcome: Change in Left Ventricular End Systolic Volume Index (LVESVI) From Randomization to 6 Months
Description: The endpoint will be a subject's change in Left Ventricular End Systolic Volume Index (a measure of the volume of blood in the left ventricle at the end of systole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 6 month - randomization visit difference in LVESVI. Negative values correspond to reductions in LVESVI over time.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 279 | 272
ml/square meter of body surface area | -6.8 (17.1) | 0.4 (17.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESVI from randomization to 6 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVESVI from randomization to 6 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESVI through 6 months was used; Posterior BiV - RV Mean Difference = -7.204, 95% CI 2-sided [-10.12 to -4.214] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESVI change through 6 months

21. Secondary Outcome: Change in Left Ventricular End Systolic Volume Index (LVESVI) From Randomization to 12 Months
Description: The endpoint will be a subject's change in Left Ventricular End Systolic Volume Index (a measure of the volume of blood in the left ventricle at the end of systole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 12 month - randomization visit difference in LVESVI. Negative values correspond to reductions in LVESVI over time.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 260 | 256
ml/square meter of body surface area | -6.8 (18.7) | 0.5 (20.2)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESVI from randomization to 12 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVESVI from randomization to 12 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESVI through 12 months was used; Posterior BiV - RV Mean Difference = -7.255, 95% CI 2-sided [-10.590 to -3.829] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESVI change through 12 months

22. Secondary Outcome: Change in Left Ventricular End Systolic Volume Index (LVESVI) From Randomization to 18 Months
Description: The endpoint will be a subject's change in Left Ventricular End Systolic Volume Index (a measure of the volume of blood in the left ventricle at the end of systole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 18 month - randomization visit difference in LVESVI. Negative values correspond to reductions in LVESVI over time.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 219 | 225
ml/square meter of body surface area | -8.8 (18.9) | -0.5 (19.9)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESVI from randomization to 18 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVESVI from randomization to 18 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESVI through 18 months was used; Posterior BiV - RV Mean Difference = -8.242, 95% CI 2-sided [-11.860 to -4.574] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESVI change through 18 months

23. Secondary Outcome: Change in Left Ventricular End Systolic Volume Index (LVESVI) From Randomization to 24 Months
Description: The endpoint will be a subject's change in Left Ventricular End Systolic Volume Index (a measure of the volume of blood in the left ventricle at the end of systole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 24 month - randomization visit difference in LVESVI. Negative values correspond to reductions in LVESVI over time.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 187 | 204
ml/square meter of body surface area | -6.0 (22.6) | 1.4 (21.3)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESVI from randomization to 24 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVESVI from randomization to 24 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESVI through 24 months was used; Posterior BiV - RV Mean Difference = -7.268, 95% CI 2-sided [-11.690 to -2.846] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESVI change through 24 months

24. Secondary Outcome: Change in Left Ventricular End Diastolic Volume Index (LVEDVI) From Randomization to 6 Months
Description: The endpoint will be a subject's change in Left Ventricular End Diastolic Volume Index (a measure of the volume of blood in the left ventricle at the end of diastole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 6 month - randomization visit difference in LVEDVI. Negative values correspond to reductions in LVEDVI over time.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 281 | 273
ml/square meter of body surface area | -6.2 (19.2) | -0.3 (19.5)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDVI from randomization to 6 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEDVI from randomization to 6 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDVI through 6 months was used; Posterior BiV - RV Mean Difference = -5.858, 95% CI 2-sided [-9.085 to -2.562] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDVI change through 6 months

25. Secondary Outcome: Change in Left Ventricular End Diastolic Volume Index (LVEDVI) From Randomization to 12 Months
Description: The endpoint will be a subject's change in Left Ventricular End Diastolic Volume Index (a measure of the volume of blood in the left ventricle at the end of diastole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 12 month - randomization visit difference in LVEDVI. Negative values correspond to reductions in LVEDVI over time.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 261 | 256
ml/square meter of body surface area | -7.0 (20.6) | -1.1 (22.2)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDVI from randomization to 12 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEDVI from randomization to 12 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDVI through 12 months was used; Posterior BiV - RV Mean Difference = -5.807, 95% CI 2-sided [-9.467 to -2.038] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDVI change through 12 months

26. Secondary Outcome: Change in Left Ventricular End Diastolic Volume Index (LVEDVI) From Randomization to 18 Months
Description: The endpoint will be a subject's change in Left Ventricular End Diastolic Volume Index (a measure of the volume of blood in the left ventricle at the end of diastole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 18 month - randomization visit difference in LVEDVI. Negative values correspond to reductions in LVEDVI over time.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 220 | 225
ml/square meter of body surface area | -9.8 (21.4) | -0.8 (22.4)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDVI from randomization to 18 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEDVI from randomization to 18 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDVI through 18 months was used; Posterior BiV - RV Mean Difference = -8.844, 95% CI 2-sided [-12.910 to -4.681] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDVI change through 18 months

27. Secondary Outcome: Change in Left Ventricular End Diastolic Volume Index (LVEDVI) From Randomization to 24 Months
Description: The endpoint will be a subject's change in Left Ventricular End Diastolic Volume Index (a measure of the volume of blood in the left ventricle at the end of diastole, normalized over body surface area). In other words, a measure of the size of the left ventricle. For each subject the measure is the 24 month - randomization visit difference in LVEDVI. Negative values correspond to reductions in LVEDVI over time.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: ml/square meter of body surface area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 189 | 206
ml/square meter of body surface area | -6.9 (24.9) | -0.1 (23.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDVI from randomization to 24 months as corresponding patients who receive right ventricular pacing. This was tested against the hypothesis that patients with biventricular pacing have a different change in LVEDVI from randomization to 24 months than patients with right ventricular pacing; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDVI through 24 months was used; Posterior BiV - RV Mean Difference = -6.615, 95% CI 2-sided [-11.370 to -1.736] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDVI change through 24 months

28. Secondary Outcome: Change in Left Ventricular Mass (LV Mass) From Randomization to 6 Months
Description: The endpoint will be a subject's change in Left Ventricular Mass ( a measure of the size of the left ventricle) from randomization to 6 months. For each subject the measurement was calculated as 6 month - randomization visit difference in LV mass measurement. Negative values correspond to a reduction in LV mass over time.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 220 | 208
grams | -8.4 (43.1) | -4.2 (47.5)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in LV Mass through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in LV Mass through 6 months with BiV pacing than RV pacing. Change was calculated as 6 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LV Mass through 6 months was used; Posterior BiV - RV Mean Difference = -3.894, 95% CI 2-sided [-12.130 to 3.953] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LV Mass change through 6 months

29. Secondary Outcome: Change in Left Ventricular Mass (LV Mass) From Randomization to 12 Months
Description: The endpoint will be a subject's change in Left Ventricular Mass ( a measure of the size of the left ventricle) from randomization to 12 months. For each subject the measurement was calculated as 12 month - randomization visit difference in LV mass measurement. Negative values correspond to a reduction in LV mass over time.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 211 | 199
grams | -15.8 (46.8) | -4.7 (52.4)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in LV Mass through 12 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in LV Mass through 12 months with BiV pacing than RV pacing. Change was calculated as 12 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LV Mass through 12 months was used; Posterior BiV - RV Mean Difference = -10.160, 95% CI 2-sided [-19.330 to -0.857] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LV Mass change through 12 months

30. Secondary Outcome: Change in Left Ventricular Mass (LV Mass) From Randomization to 18 Months
Description: The endpoint will be a subject's change in Left Ventricular Mass ( a measure of the size of the left ventricle) from randomization to 18 months. For each subject the measurement was calculated as 18 month - randomization visit difference in LV mass measurement. Negative values correspond to a reduction in LV mass over time.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 168 | 176
grams | -16.8 (48.8) | -7.2 (49.8)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in LV Mass through 18 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in LV Mass through 18 months with BiV pacing than RV pacing. Change was calculated as 18 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LV Mass through 18 months was used; Posterior BiV - RV Mean Difference = -8.316, 95% CI 2-sided [-18.190 to 1.623] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LV Mass change through 18 months

31. Secondary Outcome: Change in Left Ventricular Mass (LV Mass) From Randomization to 24 Months
Description: The endpoint will be a subject's change in Left Ventricular Mass ( a measure of the size of the left ventricle) from randomization to 24 months. For each subject the measurement was calculated as 24 month - randomization visit difference in LV mass measurement. Negative values correspond to a reduction in LV mass over time.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 150 | 163
grams | -19.4 (45.1) | -6.8 (49.6)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in LV Mass through 24 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in LV Mass through 24 months with BiV pacing than RV pacing. Change was calculated as 24 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LV Mass through 24 months was used; Posterior BiV - RV Mean Difference = -11.080, 95% CI 2-sided [-21.110 to -0.956] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LV Mass change through 24 months

32. Secondary Outcome: Change in Left Ventricular End Diastolic Dimension (LVEDD) From Randomization to 6 Months
Description: The endpoint will be a subject's change in LVEDD (a measure of the dimension of the left ventricle at the end of diastole). For each subject the measure was the 6 month - randomization visit difference in LVEDD value. Negative values correspond to reductions in LVEDD.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 254 | 242
cm | -0.1 (0.6) | 0.0 (0.6)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDD from randomization to 6 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVEDD from randomization to 6 months than patients with RV pacing. Negative values reflect reductions in LVEDD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDD through 6 months was used; Posterior BiV - RV Mean Difference = -0.126, 95% CI 2-sided [-0.235 to -0.014] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDD change through 6 months

33. Secondary Outcome: Change in Left Ventricular End Diastolic Dimension (LVEDD) From Randomization to 12 Months
Description: The endpoint will be a subject's change in LVEDD (a measure of the dimension of the left ventricle at the end of diastole). For each subject the measure was the 12 month - randomization visit difference in LVEDD value. Negative values correspond to reductions in LVEDD.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 241 | 232
cm | -0.1 (0.7) | 0.0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDD from randomization to 12 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVEDD from randomization to 12 months than patients with RV pacing. Negative values reflect reductions in LVEDD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDD through 12 months was used; Posterior BiV - RV Mean Difference = -0.162, 95% CI 2-sided [-0.287 to -0.035] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDD change through 12 months

34. Secondary Outcome: Change in Left Ventricular End Diastolic Dimension (LVEDD) From Randomization to 18 Months
Description: The endpoint will be a subject's change in LVEDD (a measure of the dimension of the left ventricle at the end of diastole). For each subject the measure was the 18 month - randomization visit difference in LVEDD value. Negative values correspond to reductions in LVEDD.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 201 | 204
cm | -0.2 (0.6) | 0.0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDD from randomization to 18 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVEDD from randomization to 18 months than patients with RV pacing. Negative values reflect reductions in LVEDD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDD through 18 months was used; Posterior BiV - RV Mean Difference = -0.163, 95% CI 2-sided [-0.293 to -0.030] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDD change through 18 months

35. Secondary Outcome: Change in Left Ventricular End Diastolic Dimension (LVEDD) From Randomization to 24 Months
Description: The endpoint will be a subject's change in LVEDD (a measure of the dimension of the left ventricle at the end of diastole). For each subject the measure was the 24 month - randomization visit difference in LVEDD value. Negative values correspond to reductions in LVEDD.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 175 | 186
cm | -0.3 (0.7) | 0.0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVEDD from randomization to 24 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVEDD from randomization to 24 months than patients with RV pacing. Negative values reflect reductions in LVEDD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVEDD through 24 months was used; Posterior BiV - RV Mean Difference = -0.245, 95% CI 2-sided [-0.390 to -0.097] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVEDD change through 24 months

36. Secondary Outcome: Change in Left Ventricular End Systolic Dimension (LVESD) From Randomization to 6 Months
Description: The endpoint will be a subject's change in LVESD (a measure of the dimension of the left ventricle at the end of systole). For each subject the measure was the 6 month - randomization visit difference in LVESD value. Negative values correspond to reductions in LVESD.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 250 | 241
cm | -0.1 (0.6) | 0.0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESD from randomization to 6 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVESD from randomization to 6 months than patients with RV pacing. Negative values reflect reductions in LVESD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESD through 6 months was used; Posterior BiV - RV Mean Difference = -0.066, 95% CI 2-sided [-0.185 to 0.055] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESD change through 6 months

37. Secondary Outcome: Change in Left Ventricular End Systolic Dimension (LVESD) From Randomization to 12 Months
Description: The endpoint will be a subject's change in LVESD (a measure of the dimension of the left ventricle at the end of systole). For each subject the measure was the 12 month - randomization visit difference in LVESD value. Negative values correspond to reductions in LVESD.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 239 | 231
cm | 0.0 (0.7) | 0.1 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESD from randomization to 12 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVESD from randomization to 12 months than patients with RV pacing. Negative values reflect reductions in LVESD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESD through 12 months was used; Posterior BiV - RV Mean Difference = -0.104, 95% CI 2-sided [-0.236 to 0.029] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESD change through 12 months

38. Secondary Outcome: Change in Left Ventricular End Systolic Dimension (LVESD) From Randomization to 18 Months
Description: The endpoint will be a subject's change in LVESD (a measure of the dimension of the left ventricle at the end of systole). For each subject the measure was the 18 month - randomization visit difference in LVESD value. Negative values correspond to reductions in LVESD.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 199 | 204
cm | -0.1 (0.7) | 0.0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESD from randomization to 18 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVESD from randomization to 18 months than patients with RV pacing. Negative values reflect reductions in LVESD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESD through 18 months was used; Posterior BiV - RV Mean Difference = -0.060, 95% CI 2-sided [-0.204 to 0.087] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESD change through 18 months

39. Secondary Outcome: Change in Left Ventricular End Systolic Dimension (LVESD) From Randomization to 24 Months
Description: The endpoint will be a subject's change in LVESD (a measure of the dimension of the left ventricle at the end of systole). For each subject the measure was the 24 month - randomization visit difference in LVESD value. Negative values correspond to reductions in LVESD.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 173 | 185
cm | -0.1 (0.8) | 0.1 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, and NYHA classifications of I, II, or III who receive biventricular pacing have the same average change in LVESD from randomization to 24 months as similar patients who receive right ventricular pacing. This was tested against the hypothesis that patients with BiV pacing have a different change in LVESD from randomization to 24 months than patients with RV pacing. Negative values reflect reductions in LVESD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in LVESD through 24 months was used; Posterior BiV - RV Mean Difference = -0.180, 95% CI 2-sided [-0.339 to -0.018] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean LVESD change through 24 months

40. Secondary Outcome: Change in Mitral Regurgitation From Randomization to 6 Months
Description: The endpoint will be a subject's change in mitral regurgitation (a measure of how much blood flows backwards into the heart due to the mitral valve not closing properly). The measure for each subject will be the 6 month - randomization visit difference in mitral regurgitation. Negative values reflect reductions in mitral regurgitation over time.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: percentage of left atrial area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 247 | 225
percentage of left atrial area | -1.3 (12.4) | -0.6 (11.2)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Mitral Regurgitation (MR) through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Mitral Regurgitation through 6 months with BiV pacing than RV pacing. Change was calculated as 6 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in MR through 6 months was used; Posterior BiV - RV Mean Difference = -0.683, 95% CI 2-sided [-2.828 to 1.506] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean MR change through 6 months

41. Secondary Outcome: Change in Mitral Regurgitation From Randomization to 12 Months
Description: The endpoint will be a subject's change in mitral regurgitation (a measure of how much blood flows backwards into the heart due to the mitral valve not closing properly). The measure for each subject will be the 12 month - randomization visit difference in mitral regurgitation. Negative values reflect reductions in mitral regurgitation over time.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: percentage of left atrial area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 235 | 214
percentage of left atrial area | -1.3 (12.0) | -0.8 (12.6)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Mitral Regurgitation (MR) through 12 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Mitral Regurgitation through 12 months with BiV pacing than RV pacing. Change was calculated as 12 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in MR through 12 months was used; Posterior BiV - RV Mean Difference = -0.564, 95% CI 2-sided [-2.843 to 1.773] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean MR change through 12 months

42. Secondary Outcome: Change in Mitral Regurgitation From Randomization to 18 Months
Description: The endpoint will be a subject's change in mitral regurgitation (a measure of how much blood flows backwards into the heart due to the mitral valve not closing properly). The measure for each subject will be the 18 month - randomization visit difference in mitral regurgitation. Negative values reflect reductions in mitral regurgitation over time.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: percentage of left atrial area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 188 | 195
percentage of left atrial area | -1.9 (12.1) | -1.9 (11.5)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Mitral Regurgitation (MR) through 18 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Mitral Regurgitation through 18 months with BiV pacing than RV pacing. Change was calculated as 18 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in MR through 18 months was used; Posterior BiV - RV Mean Difference = 0.016, 95% CI 2-sided [-2.379 to 2.425] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean MR change through 18 months

43. Secondary Outcome: Change in Mitral Regurgitation From Randomization to 24 Months
Description: The endpoint will be a subject's change in mitral regurgitation (a measure of how much blood flows backwards into the heart due to the mitral valve not closing properly). The measure for each subject will be the 24 month - randomization visit difference in mitral regurgitation. Negative values reflect reductions in mitral regurgitation over time.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: percentage of left atrial area
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 173 | 173
percentage of left atrial area | -1.1 (13.6) | -0.5 (11.4)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Mitral Regurgitation (MR) through 24 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Mitral Regurgitation through 24 months with BiV pacing than RV pacing. Change was calculated as 24 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in MR through 24 months was used; Posterior BiV - RV Mean Difference = -0.653, 95% CI 2-sided [-3.337 to 2.046] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean MR change through 24 months

44. Secondary Outcome: Change in Cardiac Index From Randomization to 6 Months
Description: The endpoint will be a subject's change in cardiac index (a measure of how much blood the left ventricle ejects in one minute, normalized over body surface area) from randomization to 6 months. The measure for each subject will be the 6 month - randomization visit value.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: liters per minute per squared meter
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 275 | 268
liters per minute per squared meter | 0 (0.6) | -0.1 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Cardiac Index (CI) through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Cardiac Index through 6 months with BiV pacing than RV pacing. Change was calculated as 6 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in CI through 6 months was used; Posterior BiV - RV Mean Difference = 0.080, 95% CI 2-sided [-0.031 to 0.195] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean CI change through 6 months

45. Secondary Outcome: Change in Cardiac Index From Randomization to 12 Months
Description: The endpoint will be a subject's change in cardiac index (a measure of how much blood the left ventricle ejects in one minute, normalized over body surface area) from randomization to 12 months. The measure for each subject will be the 12 month - randomization visit value.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: liters per minute per squared meter
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 257 | 250
liters per minute per squared meter | -0.1 (0.6) | -0.2 (0.6)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Cardiac Index (CI) through 12 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Cardiac Index through 12 months with BiV pacing than RV pacing. Change was calculated as 12 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in CI through 12 months was used; Posterior BiV - RV Mean Difference = 0.086, 95% CI 2-sided [-0.022 to 0.198] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean CI change through 12 months

46. Secondary Outcome: Change in Cardiac Index From Randomization to 18 Months
Description: The endpoint will be a subject's change in cardiac index (a measure of how much blood the left ventricle ejects in one minute, normalized over body surface area) from randomization to 18 months. The measure for each subject will be the 18 month - randomization visit value.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: liters per minute per squared meter
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 215 | 218
liters per minute per squared meter | -0.1 (0.7) | 0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Cardiac Index (CI) through 18 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Cardiac Index through 18 months with BiV pacing than RV pacing. Change was calculated as 18 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in CI through 18 months was used; Posterior BiV - RV Mean Difference = -0.081, 95% CI 2-sided [-0.218 to 0.058] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean CI change through 18 months

47. Secondary Outcome: Change in Cardiac Index From Randomization to 24 Months
Description: The endpoint will be a subject's change in cardiac index (a measure of how much blood the left ventricle ejects in one minute, normalized over body surface area) from randomization to 24 months. The measure for each subject will be the 24 month - randomization visit value.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: liters per minute per squared meter
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 186 | 198
liters per minute per squared meter | -0.1 (0.7) | -0.2 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in Cardiac Index (CI) through 24 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in Cardiac Index through 24 months with BiV pacing than RV pacing. Change was calculated as 24 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in CI through 24 months was used; Posterior BiV - RV Mean Difference = 0.047, 95% CI 2-sided [-0.095 to 0.192] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean CI change through 24 months

48. Secondary Outcome: Change in Interventricular Mechanical Delay (IVMD) From Randomization to 6 Months
Description: The endpoint will be a subject's change in interventricular mechanical delay (a measure of dyssynchrony between ventricles, measured in ms) from randomization to the 6 month visit. The measure will be the 6 month - randomization visit difference in IVMD.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 220 | 208
ms | 49.9 (134.2) | -4.2 (136.1)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in IVMD through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in IVMD through 6 months with BiV pacing than RV pacing. Change was calculated as 6 month value - randomization visit value. A positive value reflected reduction in IVMD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in IVMD through 6 months was used; Posterior BiV - RV Mean Difference = 29.300, 95% CI 2-sided [10.040 to 48.640] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean IVMD change through 6 months

49. Secondary Outcome: Change in Interventricular Mechanical Delay (IVMD) From Randomization to 12 Months
Description: The endpoint will be a subject's change in interventricular mechanical delay (a measure of dyssynchrony between ventricles, measured in ms) from randomization to the 12 month visit. The measure will be the 12 month - randomization visit difference in IVMD.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 202 | 198
ms | 38.5 (121.9) | 0.4 (128.9)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in IVMD through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in IVMD through 12 months with BiV pacing than RV pacing. Change was calculated as 12 month value - randomization visit value. A positive value reflected reduction in IVMD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in IVMD through 12 months was used; Posterior BiV - RV Mean Difference = 21.830, 95% CI 2-sided [2.841 to 40.870] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean IVMD change through 12 months

50. Secondary Outcome: Change in Interventricular Mechanical Delay (IVMD) From Randomization to 18 Months
Description: The endpoint will be a subject's change in interventricular mechanical delay (a measure of dyssynchrony between ventricles, measured in ms) from randomization to the 18 month visit. The measure will be the 18 month - randomization visit difference in IVMD.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 173 | 172
ms | 55.1 (135.7) | -0.8 (136.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in IVMD through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in IVMD through 18 months with BiV pacing than RV pacing. Change was calculated as 18 month value - randomization visit value. A positive value reflected reduction in IVMD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in IVMD through 18 months was used; Posterior BiV - RV Mean Difference = 26.530, 95% CI 2-sided [6.247 to 47.190] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean IVMD change through 18 months

51. Secondary Outcome: Change in Interventricular Mechanical Delay (IVMD) From Randomization to 24 Months
Description: The endpoint will be a subject's change in interventricular mechanical delay (a measure of dyssynchrony between ventricles, measured in ms) from randomization to the 24 month visit. The measure will be the 24 month - randomization visit difference in IVMD.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 150 | 160
ms | 48.6 (138.1) | -4.9 (133.3)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in IVMD through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in IVMD through 24 months with BiV pacing than RV pacing. Change was calculated as 24 month value - randomization visit value. A positive value reflected reduction in IVMD; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in IVMD through 24 months was used; Posterior BiV - RV Mean Difference = 23.32, 95% CI 2-sided [1.999 to 44.530] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean IVMD change through 24 months

52. Secondary Outcome: Change in E Wave/A Wave Ratio (E:A Ratio) From Randomization to 6 Months
Description: The endpoint will be a subject's change in E:A ratio (a measure of diastolic function) from randomization to 6 months. The measure for each subject will be the 6 month - randomization visit difference in E:A ratio. Typical values for the E:A ratio at a single time point are 1.04 in men and 1.03 in women.
Time Frame: Randomization to 6 Months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 221 | 194
ratio | 0 (0.6) | 0 (0.7)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in E:A ratio (E/A) through 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in E:A ratio through 6 months with BiV pacing than RV pacing. Change was calculated as 6 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in E/A through 6 months was used; Posterior BiV - RV Mean Difference = -0.047, 95% CI 2-sided [-0.180 to 0.089] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean E/A change through 6 months

53. Secondary Outcome: Change in E Wave/A Wave Ratio (E:A Ratio) From Randomization to 12 Months
Description: The endpoint will be a subject's change in E:A ratio (a measure of diastolic function) from randomization to 12 months. The measure for each subject will be the 12 month - randomization visit difference in E:A ratio. Typical values for the E:A ratio at a single time point are 1.04 in men and 1.03 in women.
Time Frame: Randomization to 12 Months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 208 | 188
ratio | 0.1 (0.7) | 0.2 (1.0)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in E:A ratio (E/A) through 12 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in E:A ratio through 12 months with BiV pacing than RV pacing. Change was calculated as 12 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in E/A through 12 months was used; Posterior BiV - RV Mean Difference = -0.117, 95% CI 2-sided [-0.287 to 0.058] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean E/A change through 12 months

54. Secondary Outcome: Change in E Wave/A Wave Ratio (E:A Ratio) From Randomization to 18 Months
Description: The endpoint will be a subject's change in E:A ratio (a measure of diastolic function) from randomization to 18 months. The measure for each subject will be the 18 month - randomization visit difference in E:A ratio. Typical values for the E:A ratio at a single time point are 1.04 in men and 1.03 in women.
Time Frame: Randomization to 18 Months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 174 | 159
ratio | 0.1 (0.8) | 0.1 (0.8)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in E:A ratio (E/A) through 18 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in E:A ratio through 18 months with BiV pacing than RV pacing. Change was calculated as 18 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in E/A through 18 months was used; Posterior BiV - RV Mean Difference = 0.041, 95% CI 2-sided [-0.136 to 0.220] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean E/A change through 18 months

55. Secondary Outcome: Change in E Wave/A Wave Ratio (E:A Ratio) From Randomization to 24 Months
Description: The endpoint will be a subject's change in E:A ratio (a measure of diastolic function) from randomization to 24 months. The measure for each subject will be the 24 month - randomization visit difference in E:A ratio. Typical values for the E:A ratio at a single time point are 1.04 in men and 1.03 in women.
Time Frame: Randomization to 24 Months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 160 | 141
ratio | 0.2 (0.8) | 0.1 (0.9)
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar changes in E:A ratio (E/A) through 24 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients have different changes in E:A ratio through 24 months with BiV pacing than RV pacing. Change was calculated as 24 month value - randomization visit value; Test type: Superiority or Other; Bayesian Credible Interval — BLOCK HF is a Bayesian study; a p-value was not used since it is a non-Bayesian statistical tool. Instead,a posterior distribution representing the set of possible values for the BiV - RV difference in change in E/A through 24 months was used; Posterior BiV - RV Mean Difference = 0.110, 95% CI 2-sided [-0.085 to 0.311] — Because Bayesian analyses were employed, a 95% two-sided credible interval was used instead of a confidence interval. This reflects the 2.5th and 97.5th percentile of possible values for the BiV-RV difference in mean E/A change through 24 months

56. Secondary Outcome: Clinical Composite Score at 6 Months
Description: The endpoint will be a subject's Clinical Composite Score at 6 months. The Clinical Composite Score is a 3 point score (Worsened, Unchanged, and Improved) based on a number of factors including: whether the subject has died, whether the subject has experienced a heart failure-related hospitalization, whether the subject has discontinued their therapy due to worsening heart failure, whether their New York Heart Association classification has improved or worsened since randomization, and whether they feel moderately or markedly better since randomization.
Time Frame: Randomization to 6 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 349 | 342
participants
  Improved | 184 | 133
  Unchanged | 83 | 113
  Worsened | 82 | 96
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar Clinical Composite Scores after 6 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients had better scores with BiV pacing than RV pacing. The analysis assigned numerical values (Improved=3, Unchanged=2, Worsened=1) and compared the average score between randomization arms using a one-sided analysis; Test type: Superiority or Other; p = 0.9985, Posterior probability of mean difference — BLOCK HF is a Bayesian study; a p-value was not used. Instead, a posterior probability, representing the probability that subjects with biventricular pacing have better outcomes, was calculated. A probability ≥ 0.95 was significant; The posterior probability that the mean difference is greater than 0 was calculated; Mean Difference (Final Values) = 0.1841 — This was a one-sided analysis of the BiV arm - RV arm difference in Mean Clinical Composite Scores. Values above 0 suggested better outcomes in the Biventricular arm

57. Secondary Outcome: Clinical Composite Score at 12 Months
Description: The endpoint will be a subject's Clinical Composite Score at 12 months. The Clinical Composite Score is a 3 point score (Worsened, Unchanged, and Improved) based on a number of factors including: whether the subject has died, whether the subject has experienced a heart failure-related hospitalization, whether the subject has discontinued their therapy due to worsening heart failure, whether their New York Heart Association classification has improved or worsened since randomization, and whether they feel moderately or markedly better since randomization.
Time Frame: Randomization to 12 Months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Biventricular Pacing Arm: Subjects randomized to receive biventricular pacing who either worsened prior to the 12 month visit or did not miss their 12 month visit due to study closure
- Right Ventricular Pacing Arm: Subjects randomized to receive right ventricular pacing who either worsened prior to the 12 month visit or did not miss their 12 month visit due to study closure
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 345 | 341
participants
  Improved | 160 | 117
  Unchanged | 82 | 78
  Worsened | 103 | 146
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar Clinical Composite Scores after 12 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients had better scores with BiV pacing than RV pacing. The analysis assigned numerical values (Improved=3, Unchanged=2, Worsened=1) and compared the average score between randomization arms using a one-sided analysis; Test type: Superiority or Other; p = 0.9999, Posterior probability of mean difference — [p-value comment as in outcome 56, analysis 1]; The posterior probability that the mean difference is greater than 0 was calculated; Mean Difference (Final Values) = 0.2503 — [estimate comment as in outcome 56, analysis 1]

58. Secondary Outcome: Clinical Composite Score at 18 Months
Description: The endpoint will be a subject's Clinical Composite Score at 18 months. The Clinical Composite Score is a 3 point score (Worsened, Unchanged, and Improved) based on a number of factors including: whether the subject has died, whether the subject has experienced a heart failure-related hospitalization, whether the subject has discontinued their therapy due to worsening heart failure, whether their New York Heart Association classification has improved or worsened since randomization, and whether they feel moderately or markedly better since randomization.
Time Frame: Randomization to 18 Months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Biventricular Pacing Arm: Subjects randomized to receive biventricular pacing who either worsened prior to the 18 month visit or did not miss their 18 month visit due to study closure
- Right Ventricular Pacing Arm: Subjects randomized to receive right ventricular pacing who either worsened prior to the 18 month visit or did not miss their 18 month visit due to study closure
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 325 | 323
participants
  Improved | 137 | 103
  Unchanged | 68 | 70
  Worsened | 120 | 150
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar Clinical Composite Scores after 18 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients had better scores with BiV pacing than RV pacing. The analysis assigned numerical values (Improved=3, Unchanged=2, Worsened=1) and compared the average score between randomization arms using a one-sided analysis; Test type: Superiority or Other; p = 0.9978, Posterior probability of mean difference — [p-value comment as in outcome 56, analysis 1]; The posterior probability that the mean difference is greater than 0 was calculated; Mean Difference (Final Values) = 0.1978 — [estimate comment as in outcome 56, analysis 1]

59. Secondary Outcome: Clinical Composite Score at 24 Months
Description: The endpoint will be a subject's Clinical Composite Score at 24 months. The Clinical Composite Score is a 3 point score (Worsened, Unchanged, and Improved) based on a number of factors including: whether the subject has died, whether the subject has experienced a heart failure-related hospitalization, whether the subject has discontinued their therapy due to worsening heart failure, whether their New York Heart Association classification has improved or worsened since randomization, and whether they feel moderately or markedly better since randomization.
Time Frame: Randomization to 24 Months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Biventricular Pacing Arm: Subjects randomized to receive biventricular pacing who either worsened prior to the 24 month visit or did not miss their 24 month visit due to study closure
- Right Ventricular Pacing Arm: Subjects randomized to receive right ventricular pacing who either worsened prior to the 24 month visit or did not miss their 24 month visit due to study closure
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm
Number analyzed (Participants) | 308 | 314
participants
  Improved | 118 | 94
  Unchanged | 70 | 59
  Worsened | 120 | 161
Statistical Analysis 1: Comparison: Biventricular Pacing Arm vs Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, NYHA I-III, and LVEF of at most 50% who receive RV pacing have similar Clinical Composite Scores after 24 months compared to similar patients who receive BiV pacing. This was tested against the alternative hypothesis that patients had better scores with BiV pacing than RV pacing. The analysis assigned numerical values (Improved=3, Unchanged=2, Worsened=1) and compared the average score between randomization arms using a one-sided analysis; Test type: Superiority or Other; p = 0.9983, Posterior probability of mean difference — [p-value comment as in outcome 56, analysis 1]; The posterior probability that the mean difference is greater than 0 was calculated; Mean Difference (Final Values) = 0.2069 — [estimate comment as in outcome 56, analysis 1]

60. Secondary Outcome: CRT-P and CRT-D System Implant Success
Description: The endpoint will be whether each subject who underwent an implant attempt of a Cardiac Resynchronization Therapy device, be it a pacing only device (CRT-P) or a pacing device with defibrillation capability (CRT-D), had a successful procedure (i.e. the generator, left ventricular lead, and right ventricular lead were successfully implanted). Only one implant attempt was allowed.
Time Frame: Initial Implant Procedure
Population: For this outcome measure, only subjects in the "No Implant Attempt" subgroup were excluded.
Measure: Number; unit: participants
Groups:
- Subjects With a CRT-P Implant Attempt: Subjects who underwent an implant attempt for a CRT-P device
- Subjects With a CRT-D Implant Attempt: Subjects who underwent an implant attempt for a CRT-D device
Arm/Group | Subjects With a CRT-P Implant Attempt | Subjects With a CRT-D Implant Attempt
Number analyzed (Participants) | 561 | 248
participants
  Subjects successfully implanted | 531 | 227
  Subjects not successfully implanted | 30 | 21

61. Secondary Outcome: Incidence of Ventricular Tachyarrhythmias
Description: Among subjects implanted with a Cardiac Resynchronization Therapy with Defibrillation device (CRT-D) and randomized, the endpoint was the time from randomization until the subject experienced a ventricular tachyarrhythmia. For each randomization arm, the number of CRT-D subjects who experienced at least one ventricular tachyarrhythmia post-randomization is reported, as well as the number of CRT-D subjects who did not experience one or more ventricular tachyarrhythmias post-randomization.
Time Frame: Participants were followed for the duration of the study, an average of 37.9 months post-randomization among CRT-D subjects.
Population: Only randomized subjects in the CRT-D device group were included in the analysis of this endpoint, as the analysis was restricted to post-randomization data recorded by CRT-D devices. Subjects in the "No Implant Attempt", "Unsuccessful Implants", "CRT-D: Not Randomized", and all CRT-P subgroups were excluded.
Measure: Number; unit: participants
Arm/Group | CRT-D: Biventricular Pacing Arm | CRT-D: Right Ventricular Pacing Arm
Number analyzed (Participants) | 106 | 101
participants
  Subjects who experienced VT/VF | 39 | 31
  Subjects who did not experience VT/VF | 67 | 70
Statistical Analysis 1: Comparison: CRT-D: Biventricular Pacing Arm vs CRT-D: Right Ventricular Pacing Arm; The null hypothesis is that patients with AV block, ejection fractions of at most 50%, NYHA classifications of I-III, and indicated for defibrillation therapy who receive biventricular (BiV) pacing have the same rate of experiencing their first ventricular arrhythmia as corresponding patients who receive right ventricular pacing. This was tested against the one-side hypothesis that patients with BiV pacing have a lower risk of ventricular arrhythmias than subjects with right ventricular pacing; Test type: Superiority or Other; p = 0.189, Posterior Distribution for HR — BLOCK HF is a Bayesian study; a p-value was not used. Instead, a posterior probability, representing the probability that subjects with biventricular pacing have better outcomes, were calculated. A probability ≥ 0.95 was significant; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.78 to 2.01] — The hazard ratio corresponds to the time from randomization to first ventricular arrhythmia occurring post-randomization for each subject. Ventricular arrhythmias occurring prior to randomization were excluded. A 95% credible interval was used

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after the date of consent and on or before the date of exit
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE. In the case of the BiV and RV randomized arms, both pre-randomization and post-randomization adverse events are included.
Groups:
- Biventricular Pacing Arm: Subjects who were implanted with a CRT device and randomized to receive biventricular pacing
- Right Ventricular Pacing Arm: Subjects who were implanted with a CRT device and randomized to receive right ventricular pacing
- CRT: Not Randomized: Subjects successfully implanted with a CRT device who were not randomized
Arm/Group | Biventricular Pacing Arm | Right Ventricular Pacing Arm | CRT: Not Randomized | Unsuccessful Implants | No Implant Attempt
Serious Adverse Events (participants affected / at risk) | 223/349 | 219/342 | 41/67 | 6/51 | 2/109
Other Adverse Events (participants affected / at risk) | 193/349 | 181/342 | 16/67 | 8/51 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biventricular Pacing Arm (N=349) | Right Ventricular Pacing Arm (N=342) | CRT: Not Randomized (N=67) | Unsuccessful Implants (N=51) | No Implant Attempt (N=109)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 8 (11) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 9 (10) | 10 (11) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 5 (7) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 14 (19) | 26 (37) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 4 (6) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (5) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 100 (196) | 117 (215) | 20 (28) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 10 (10) | 6 (7) | 1 (2) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 5 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 11 (17) | 14 (20) | 1 (3) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 5 (5) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Implant site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 28 (57) | 37 (50) | 6 (8) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (9) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication of device insertion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defibrillation threshold increased (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device lead damage (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Device migration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dialysis device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated pacing threshold (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to capture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lead dislodgement (Injury, poisoning and procedural complications) | 12 (13) | 13 (15) | 3 (3) | 3 (3) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oversensing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 14 (16) | 13 (14) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 10 (12) | 14 (16) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 8 (9) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis glandularis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 18 (20) | 15 (17) | 3 (4) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 11 (17) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device change (Surgical and medical procedures) | 39 (39) | 23 (24) | 3 (3) | 0 (0) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 8 (8) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biventricular Pacing Arm (N=349) | Right Ventricular Pacing Arm (N=342) | CRT: Not Randomized (N=67) | Unsuccessful Implants (N=51) | No Implant Attempt (N=109)
Atrial fibrillation (Cardiac disorders) | 38 (42) | 33 (36) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 63 (90) | 77 (114) | 2 (2) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 25 (30) | 20 (23) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 19 (22) | 24 (27) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 12 (13) | 17 (17) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 17 (20) | 23 (27) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (41) | 23 (32) | 5 (6) | 0 (0) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 53 (70) | 14 (14) | 5 (6) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 12 (14) | 19 (22) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 12 (12) | 26 (27) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 29 (30) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No